CLINICAL TRIAL: NCT04570150
Title: Optimizing Post-operative Recovery in Bariatric Patients With Obstructive Sleep Apnea Undergoing Outpatient Surgery: A Comparison of Sugammadex and Neostigmine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jerry Ingrande, Associate Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MISP 59701
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Active Comparator)
  Interventions: Drug: Sugammadex
- Neostigmine (Placebo Comparator)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Subjects who are randomized to into the sugammadex arm (Arm I) will receive sugammadex for reversal of neuromuscular block at the completion of their anesthetic; Outcomes measures will be recorded and compared with those from Arm II (neostigmine group).
  Arms: Sugammadex
Drug: Neostigmine — Subjects who are randomized into the neostigmine arm (Arm II) will receive neostigmine for reversal of neuromuscular block at the completion of their anesthetic; Outcomes measures will be recorded and compared with those from Arm I (sugammadex group).
  Arms: Neostigmine

SUMMARY:
This study assesses the efficacy of sugammadex against neostigmine for hastening recovery from neuromuscular blockade and optimizing pulmonary function in obese patients with obstructive sleep apnea presenting for outpatient surgery. Both drugs are used in anesthesiology to reverse neuromuscular blockade that is given in the setting of inducing and maintaining general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* obese (body mass index [BMI] >30 kg/m2)
* diagnosis of obstructive sleep apnea (OSA) (with or without continuous positive airway pressure [CPAP] use)
* scheduled for surgery requiring general anesthesia and neuromuscular blockade

Exclusion Criteria:

* history of hepatic, renal, or cardiovascular and/or cerebrovascular dysfunction
* history of difficult tracheal intubation
* history of adverse reaction to anesthesia
* history of adverse reaction to rocuronium, sugammadex, and/or neostigmine/glycopyrrolate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 8 | 6 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [38 to 61] | 49 [38 to 60] | 49 [38 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 13 | 15 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Time to PACU Discharge
Description: Time it takes from admittance to discharge from PACU.
Time Frame: Time to PACU discharge will begin at the time each subject is admitted to the PACU. The time will end immediately once the subject leaves the PACU up to a period of 300 minutes. The outcome will be measured for each subject on the day of surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 45 | 45
minutes | 123 [94 to 169] | 125 [73 to 186]

2. Secondary Outcome: Compare Proportional Changes Between Baseline Peak Expiratory Flow Rates and Postoperative Peak Expiratory Flow Rates Between Subjects Receiving Sugammadex and Those Receiving Neostigmine.
Description: Baseline peak expiratory flow rates will be measured preoperatively (units: L/min). These values will be compared with postoperative peak expiratory flow rates. The proportional change (values between 0 and 1) will be compared between subjects receiving sugammadex and subjects receiving neostigmine.
Time Frame: Baseline peak expiratory flow (PEF) will be measured 10 minutes prior to entry to the operating room; post-operative PEF will be measured 30 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: median proportional change from baseline
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 44 | 40
median proportional change from baseline | 0.57 [0.32 to 0.88] | 0.65 [0.47 to 0.91]

3. Secondary Outcome: Compare Proportional Changes Between Baseline Peak Forced Expiratory Volume Over 1 Second (FEV1) and Postoperative FEV1 Between Subjects Receiving Sugammadex and Those Receiving Neostigmine.
Description: Baseline FEV1 will be measured preoperatively (units: liters). These values will be compared with postoperative FEV1. The proportional change (values between 0 and 1) will be compared between subjects receiving sugammadex and subjects receiving neostigmine.
Time Frame: Baseline forced expiratory volume (FEV1) will be measured 10 minutes prior to entry to the operating room; post-operative FEV1 will be measured 30 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: median proportional change from baseline
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 44 | 40
median proportional change from baseline | 0.63 [0.34 to 0.88] | 0.73 [0.52 to 0.87]

4. Secondary Outcome: Compare Proportional Changes Between Baseline Forced Vital Capacity (FVC) and Postoperative FVC Between Subjects Receiving Sugammadex and Those Receiving Neostigmine.
Description: Baseline forced vital capacity (FVC) measurements will be measured preoperatively (units: Liters). These values will be compared with FVC measurements. The proportional change (values between 0 and 1) will be compared between subjects receiving sugammadex and subjects receiving neostigmine.
Time Frame: Baseline forced vital capacity (FVC) will be measured 10 minutes prior to entry to the operating room; post-operative FVC will be measured 30 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: median proportional change from baseline
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 44 | 40
median proportional change from baseline | 0.62 [0.43 to 0.93] | 0.72 [0.53 to 0.94]

5. Secondary Outcome: Compare Proportional Changes Between Baseline PaO2 Measured Via Arterial Blood Gas and Postoperative PaO2 (Measured Via Arterial Blood Gas) Between Subjects Receiving Sugammadex and Those Receiving Neostigmine.
Description: Baseline PaO2 will be measured preoperatively via an arterial blood gas (units: mmHg). These values will be compared with postoperative PaO2 values also measured via an arterial blood gas. The proportional change (values between 0 and 1) will be compared between subjects receiving sugammadex and subjects receiving neostigmine.
Time Frame: Baseline PaO2 arterial blood gas measurements will be measured 10 minutes prior to entry to the operating room; post-operative PaO2 arterial blood gas measurements will be measured 30 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: median proportional change from baseline
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 24 | 21
median proportional change from baseline | 0.74 [0.6 to 0.91] | 0.9 [0.66 to 1.13]

6. Secondary Outcome: Compare Proportional Changes Between Baseline PaCO2 Measured Via Arterial Blood Gas and Postoperative PaCO2 (Measured Via Arterial Blood Gas) Between Subjects Receiving Sugammadex and Those Receiving Neostigmine.
Description: Baseline PaCO2 will be measured preoperatively via an arterial blood gas (units: mmHg). These values will be compared with postoperative PaCO2 values also measured via an arterial blood gas. The proportional change (values between 0 and 1) will be compared between subjects receiving sugammadex and subjects receiving neostigmine.
Time Frame: Baseline PaCO2 arterial blood gas measurements will be measured 10 minutes prior to entry to the operating room; post-operative PaCO2 arterial blood gas measurements will be measured 30 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: median proportional change from baseline
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 24 | 21
median proportional change from baseline | 1.08 [0.96 to 1.18] | 1.07 [0.95 to 1.13]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Sugammadex | Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT04570150/Prot_SAP_001.pdf